CLINICAL TRIAL: NCT02603952
Title: A Phase 2a, Randomized, Partial Double-blind, Single Dose, Active-controlled, Dose Ranging Study to Evaluate the Safety of MEDI8852 in Adults With Acute, Uncomplicated Influenza
Brief Title: A Phase 2a to Evaluate the Safety of MEDI8852 in Adults With Uncomplicated Influenza
Acronym: MEDI8852
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D6000C00002
Record Dates: First submitted 2015-11-02; First posted 2015-11-13 (Estimated); Results first posted 2018-06-08 (Actual); Last update posted 2018-06-08 (Actual); Status verified 2018-05

CONDITIONS: Influenza
Keywords: Influenza; Influenza A; Flu; Flu A
MeSH Terms: conditions — Influenza, Human | interventions — Oseltamivir; MEDI8852

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo + Oseltamivir 75 mg (Placebo Comparator): Participants will receive a single intravenous (IV) infusion of placebo (matched to MEDI8852) on Day 1 and oseltamivir 75 milligrams (mg) capsules orally twice a day (BID) from Day 1 to Day 5.
  Interventions: Drug: Oseltamivir; Drug: Placebo
- MEDI8852 750 mg + Oseltamivir 75 mg (Experimental): Participants will receive a single IV infusion of MEDI8852 750 mg on Day 1 and oseltamivir 75 mg capsules orally BID from Day 1 to Day 5.
  Interventions: Drug: Oseltamivir; Drug: MEDI8852
- MEDI8852 3000 mg + Oseltamivir 75 mg (Experimental): Participants will receive a single IV infusion of MEDI8852 3000 mg on Day 1 and oseltamivir 75 mg capsules orally BID from Day 1 to Day 5.
  Interventions: Drug: Oseltamivir; Drug: MEDI8852
- MEDI8852 3000 mg (Experimental): Participants will receive a single IV infusion of MEDI8852 3000 mg on Day 1.
  Interventions: Drug: MEDI8852

INTERVENTIONS:
Drug: Oseltamivir — 75 mg capsules orally BID from Day 1 to Day 5.
  Arms: MEDI8852 3000 mg + Oseltamivir 75 mg; MEDI8852 750 mg + Oseltamivir 75 mg; Placebo + Oseltamivir 75 mg
Drug: MEDI8852 — MEDI8852 is a human IgG1 kappa monoclonal antibody (mAb) administered as a single IV infusion of 750 mg or 3000 mg on Day 1.
  Arms: MEDI8852 3000 mg; MEDI8852 3000 mg + Oseltamivir 75 mg; MEDI8852 750 mg + Oseltamivir 75 mg
Drug: Placebo — Placebo is salt-water solution containing no active ingredients and administered as a single IV infusion on Day 1.
  Arms: Placebo + Oseltamivir 75 mg

SUMMARY:
The purpose of this study is to evaluate safety and tolerability of a single dose of MEDI8852 when given with oseltamivir, the safety and tolerability of oseltamivir alone, and the safety and tolerability of a single dose of MEDI8852 alone in adult participants with acute, uncomplicated influenza caused by Type A strains.

DETAILED DESCRIPTION:
The MEDI8852 phase 2a study will evaluate the safety and tolerability of a single intravenous (IV) dose of MEDI8852 administered in conjunction with oseltamivir, the safety and tolerability of oseltamivir alone and the safety and tolerability of a single IV dose of MEDI8852 alone in adult participants with confirmed acute, uncomplicated influenza caused by Type A strains. Enrollment is planned in the United States, South Africa, and Australia.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 through 65 years at the time of screening.
* Symptomatic presumptive Influenza A infection with onset of symptoms less than or equal to (≤) 5 days prior to MEDI8852 administration and defined as the presence of:
* Fever of greater than or equal to (≥) 38.0 degrees Celsius (100.4 degrees Fahrenheit) at screening AND
* ≥ 1 moderate systemic symptom (headache, malaise, myalgia, sweats and/or chills, or fatigue) AND
* ≥ 1 moderate respiratory symptom (cough, sore throat, or nasal symptoms)
* Influenza A infection confirmed with positive rapid antigen test
* Able to complete the follow-up period through Day 101 as required by protocol (including telephone follow-up for Days 11 to 101)
* Females of childbearing potential who are sexually active with a nonsterilized male partner must use a highly effective method of contraception for at least 2 days prior to the first dose of investigational product and must agree to continue using such precautions through Day 101 of the study

Exclusion Criteria:

* Hospitalized subjects.
* Receipt of influenza antiviral therapy within the preceding 14 days.
* Receipt of immunoglobulin or blood products within 6 months prior to screening.
* Known immunodeficiency due to illness, including human immunodeficiency virus (HIV), or due to drugs, including any course of glucocorticoid therapy exceeding 2 weeks of prednisone or equivalent at a dose of 20 mg daily or every other day within 6 months prior to screening.
* Current clinical evidence of pneumonia.
* Active bacterial infection requiring treatment with oral or parenteral antibiotics.
* History of malignancy other than treated non-melanoma skin cancers or locally-treated cervical cancer in previous 3 years.
* Any planned surgical procedure before completion of Day 101.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2015-12-07 (Actual); Primary Completion 2016-12-09 (Actual); Study Completion 2016-12-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (24):
- United States (18):
  - Research Site, Canoga Park, California
  - Research Site, Long Beach, California
  - Research Site, Los Angeles, California
  - Research Site, Upland, California
  - Research Site, Hialeah, Florida
  - Research Site, Miami, Florida
  - Research Site, Miami Lakes, Florida
  - Research Site, North Miami Beach, Florida
  - Research Site, Avon, Indiana
  - Research Site, Muncie, Indiana
  - Research Site, New Orleans, Louisiana
  - Research Site, Troy, Michigan
  - Research Site, Butte, Montana
  - Research Site, Hickory, North Carolina
  - Research Site, Shelby, North Carolina
  - Research Site, Smithfield, Pennsylvania
  - Research Site, San Antonio, Texas
  - Research Site, Clinton, Utah
- South Africa (6):
  - Research Site, Durban
  - Research Site, Johannesburg
  - Research Site, Pretoria
  - Research Site, Thabazimbi
  - Research Site, Welkom
  - Research Site, Winnie Mandela

REFERENCES:
- [Derived] Ali SO, Takas T, Nyborg A, Shoemaker K, Kallewaard NL, Chiong R, Dubovsky F, Mallory RM. Evaluation of MEDI8852, an Anti-Influenza A Monoclonal Antibody, in Treating Acute Uncomplicated Influenza. Antimicrob Agents Chemother. 2018 Oct 24;62(11):e00694-18. doi: 10.1128/AAC.00694-18. Print 2018 Nov. PMID 30150460

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted from 07 Dec 2015 to 09 Dec 2016 in Australia, South Africa and United States of America.
Pre-assignment Details: A total of 373 participants were screened, of which 247 participants were screen failures and 126 participants were randomized in the study.
Groups:
- Placebo + Oseltamivir 75 mg: Participants received a single intravenous (IV) infusion of placebo (matched to MEDI8852) on Day 1 and oseltamivir 75 milligrams (mg) capsules orally twice a day (BID) from Day 1 to Day 5.
- MEDI8852 750 mg + Oseltamivir 75 mg: Participants received a single IV infusion of MEDI8852 750 mg on Day 1 and oseltamivir 75 mg capsules orally BID from Day 1 to Day 5.
- MEDI8852 3000 mg + Oseltamivir 75 mg: Participants received a single IV infusion of MEDI8852 3000 mg on Day 1 and oseltamivir 75 mg capsules orally BID from Day 1 to Day 5.
- MEDI8852 3000 mg: Participants received a single IV infusion of MEDI8852 3000 mg on Day 1.
Period: Overall Study
Arm/Group | Placebo + Oseltamivir 75 mg | MEDI8852 750 mg + Oseltamivir 75 mg | MEDI8852 3000 mg + Oseltamivir 75 mg | MEDI8852 3000 mg
Started | 32 | 31 | 31 | 32
Treated | 32 | 31 | 31 | 31
Completed | 31 | 31 | 31 | 31
Not Completed | 1 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Not completed — Received oseltamivir by error | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat population included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo + Oseltamivir 75 mg | MEDI8852 750 mg + Oseltamivir 75 mg | MEDI8852 3000 mg + Oseltamivir 75 mg | MEDI8852 3000 mg | Total
Number analyzed (Participants) | 32 | 31 | 31 | 32 | 126
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.3 (11.97) | 40.5 (11.97) | 41.7 (12.90) | 44.3 (13.96) | 42.2 (12.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 13 | 18 | 15 | 66
  Male | 12 | 18 | 13 | 17 | 60
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 17 | 20 | 17 | 70
  Not Hispanic or Latino | 16 | 14 | 11 | 15 | 56
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 5 | 8 | 3 | 5 | 21
  White | 26 | 23 | 28 | 27 | 104
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Solicited Influenza Symptoms From Day 1 Through Day 10
Description: Solicited influenza symptoms included cough, nasal congestion, sore throat, aches and pains, fatigue (tiredness), headache, chills/sweats (feeling feverish).
Time Frame: Day 1 (post-dose) through Day 10
Population: As-treated population included all participants who were randomized and received any portion of their protocol-specified treatment regimen.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + Oseltamivir 75 mg | MEDI8852 750 mg + Oseltamivir 75 mg | MEDI8852 3000 mg + Oseltamivir 75 mg | MEDI8852 3000 mg
Number analyzed (Participants) | 32 | 31 | 31 | 31
Participants
  Any symptom | 32 | 31 | 31 | 31

2. Primary Outcome: Number of Participants With Any Solicited Influenza Symptoms From Day 10 Through Day 13
Description: as for outcome 1
Time Frame: Day 10 through Day 13
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + Oseltamivir 75 mg | MEDI8852 750 mg + Oseltamivir 75 mg | MEDI8852 3000 mg + Oseltamivir 75 mg | MEDI8852 3000 mg
Number analyzed (Participants) | 32 | 31 | 31 | 31
Participants
  Any symptom | 11 | 14 | 18 | 11

3. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is any untoward medical occurrence attributed to study drug in a participant who received study drug. Treatment-emergent events were between administration of study drug and Day 28 that were absent before treatment or that worsened relative to pre-treatment state.
Time Frame: Day 1 (post-dose) through Day 28
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + Oseltamivir 75 mg | MEDI8852 750 mg + Oseltamivir 75 mg | MEDI8852 3000 mg + Oseltamivir 75 mg | MEDI8852 3000 mg
Number analyzed (Participants) | 32 | 31 | 31 | 31
Participants | 9 | 11 | 15 | 12

4. Primary Outcome: Number of Participants With Treatment-Emergent Serious Adverse Events (TESAEs)
Description: A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent events were between administration of study drug and Day 101 that were absent before treatment or that worsened relative to pre-treatment state.
Time Frame: Day 1 (post-dose) through Day 101
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + Oseltamivir 75 mg | MEDI8852 750 mg + Oseltamivir 75 mg | MEDI8852 3000 mg + Oseltamivir 75 mg | MEDI8852 3000 mg
Number analyzed (Participants) | 32 | 31 | 31 | 31
Participants | 1 | 0 | 1 | 0

5. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events of Special Interest (TEAESIs)
Description: An AE is any untoward medical occurrence attributed to study drug in a participant who received study drug. An AESI was one of scientific and medical interest specific to understanding of the study drug and may have required close monitoring and rapid communication by the investigator to the sponsor. Treatment-emergent events were between administration of study drug and Day 101 that were absent before treatment or that worsened relative to pre treatment state.
Time Frame: Day 1 (post-dose) through Day 101
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + Oseltamivir 75 mg | MEDI8852 750 mg + Oseltamivir 75 mg | MEDI8852 3000 mg + Oseltamivir 75 mg | MEDI8852 3000 mg
Number analyzed (Participants) | 32 | 31 | 31 | 31
Participants | 0 | 0 | 1 | 0

6. Secondary Outcome: Percentage of Participants With Influenza Viral Shedding as Measured by Quantitative Reverse Transcription-Polymerase Chain Reaction (qRT-PCR)
Description: Quantitative real-time polymerase chain reaction (qRT-PCR) was used to measure influenza viral shedding from the nasopharyngeal swabs. Percentage of participants who shed influenza virus are reported.
Time Frame: Baseline (Day 1) and Days 3, 5, 7, 9, 11, and 13
Population: Per-protocol (PP) population included all randomized participants who received any portion of their protocol-specified treatment regimen with valid assay results from nasopharyngeal specimens obtained at any post-dosing time point. Participants without confirmed influenza A at baseline were excluded from the PP population.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo + Oseltamivir 75 mg | MEDI8852 750 mg + Oseltamivir 75 mg | MEDI8852 3000 mg + Oseltamivir 75 mg | MEDI8852 3000 mg
Number analyzed (Participants) | 30 | 27 | 23 | 24
Percentage of Participants
  Baseline (Day 1) | 100 [88.4 to 100] | 100 [87.2 to 100] | 100 [85.2 to 100] | 100 [85.8 to 100]
  Day 3 | 90 [73.5 to 97.9] | 88.9 [70.8 to 97.6] | 91.3 [72.0 to 98.9] | 95.8 [78.9 to 99.9]
  Day 5 | 56.7 [37.4 to 74.5] | 85.2 [66.3 to 95.8] | 60.9 [38.5 to 80.3] | 54.2 [32.8 to 74.4]
  Day 7 | 33.3 [17.3 to 52.8] | 59.3 [38.8 to 77.6] | 30.4 [13.2 to 52.9] | 37.5 [18.8 to 59.4]
  Day 9 | 3.3 [0.1 to 17.2] | 7.4 [0.9 to 24.3] | 4.3 [0.1 to 21.9] | 0.0 [0.0 to 14.2]
  Day 11 | 0.0 [0.0 to 11.6] | 0.0 [0.0 to 12.8] | 0.0 [0.0 to 14.8] | 4.2 [0.1 to 21.1]
  Day 13 | 0.0 [0.0 to 11.6] | 0.0 [0.0 to 12.8] | 0.0 [0.0 to 14.8] | 0.0 [0.0 to 14.2]

7. Secondary Outcome: Quantitation of Influenza Viral Shedding as Measured by qRT-PCR
Description: qRT-PCR was used to measure influenza viral shedding from the nasopharyngeal swabs.
Time Frame: Baseline (Day 1) and Days 3, 5, 7, 9, 11, and 13
Population: PP population included all randomized participants who received any portion of their protocol-specified treatment regimen with valid assay results from nasopharyngeal specimens obtained at any post-dosing time point. Participants without confirmed influenza A at baseline were excluded from the PP population.
Measure: Mean (Standard Deviation); unit: Log10 (viral copies/mL)
Arm/Group | Placebo + Oseltamivir 75 mg | MEDI8852 750 mg + Oseltamivir 75 mg | MEDI8852 3000 mg + Oseltamivir 75 mg | MEDI8852 3000 mg
Number analyzed (Participants) | 30 | 27 | 23 | 24
Log10 (viral copies/mL)
  Baseline (Day 1) | 6.37 (1.52) | 6.62 (1.30) | 6.92 (1.17) | 6.34 (1.47)
  Day 3: number analyzed (Participants) | 29 | 27 | 22 | 23
  Day 3 | 4.35 (1.36) | 4.75 (1.31) | 4.89 (1.39) | 4.63 (1.33)
  Day 5: number analyzed (Participants) | 28 | 27 | 21 | 24
  Day 5 | 3.45 (1.03) | 3.31 (0.73) | 3.43 (1.22) | 3.73 (1.23)
  Day 7: number analyzed (Participants) | 30 | 27 | 22 | 23
  Day 7 | 2.94 (0.47) | 3.13 (0.93) | 2.97 (0.71) | 3.03 (0.57)
  Day 9: number analyzed (Participants) | 7 | 6 | 3 | 7
  Day 9 | 3.12 (0.85) | 3.76 (1.60) | 2.80 (0.00) | 2.80 (0.00)
  Day 11: number analyzed (Participants) | 3 | 2 | 3 | 4
  Day 11 | 2.80 (0.00) | 2.80 (0.00) | 2.80 (0.00) | 3.11 (0.63)
  Day 13: number analyzed (Participants) | 0 | 0 | 0 | 1
  Day 13 |  |  |  | 2.80 (NA) — Standard deviation (SD) data not applicable as only one participant was evaluable for this time point.

8. Secondary Outcome: Number of Days of Influenza Viral Shedding as Measured by qRT-PCR
Description: Number of days of viral shedding for participants who shed influenza virus is reported. qRT-PCR was used to measure influenza viral shedding from the nasopharyngeal swabs.
Time Frame: From Baseline (Day 1) to Day 7; and Day 9 to Day 13
Population: PP population. Participants without confirmed influenza A at baseline were excluded from the PP population. Participants with shedding data available for Day 1 to Day 7 and Day 9 to Day 13 were analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Placebo + Oseltamivir 75 mg | MEDI8852 750 mg + Oseltamivir 75 mg | MEDI8852 3000 mg + Oseltamivir 75 mg | MEDI8852 3000 mg
Number analyzed (Participants) | 30 | 27 | 23 | 24
Days
  Day 1 to Day 7: number analyzed (Participants) | 23 | 19 | 17 | 16
  Day 1 to Day 7 | 4.7 (2.05) | 5.8 (1.84) | 4.9 (1.95) | 4.8 (2.18)
  Day 9 to Day 13: number analyzed (Participants) | 7 | 8 | 6 | 8
  Day 9 to Day 13 | 5.4 (2.94) | 6.3 (2.60) | 6.0 (2.45) | 5.5 (2.78)

9. Secondary Outcome: Percentage of Participants With Amino Acid Changes in MEDI8852 Binding Site
Description: Genotypic analysis was performed to identify all amino acid changes in MEDI8852 binding site between each baseline (Day1) sample and the participant's corresponding last sample sequenced. Percentage of participants with changes in the amino acid corresponding to MEDI8852 binding site is reported. Due to the fact that the percentage of participants with amino acid changes in MEDI8852 binding site was zero across all participant samples analyzed, no additional per arm analyses were performed.
Time Frame: From Baseline (Day 1) to Day 13
Population: PP population. Participants without confirmed influenza A at baseline were excluded from the PP population. Participants with confirmed Influenza A positive and Influenza A concentrations greater than the lower limit of quantification (LLOQ) were analyzed.
Measure: Number; unit: Percentage of Participants
Groups:
- All MEDI8852 Participants: Participants who received a single IV infusion of MEDI8852 750 mg on Day 1 and oseltamivir 75 mg capsules orally BID from Day 1 to Day 5; or a single IV infusion of MEDI8852 3,000 mg on Day 1 and oseltamivir 75 mg capsules orally BID from Day 1 to Day 5; or a single IV infusion of MEDI8852 3000 mg on Day 1.
Arm/Group | All MEDI8852 Participants
Number analyzed (Participants) | 94
Percentage of Participants | 0

10. Secondary Outcome: Number of Participants With Viral Susceptibility to MEDI8852 as Determined by a Cell Based Microneutralization Assay
Description: Viral susceptibility to MEDI8852 was measured by a Madin-Darby canine kidney (MDCK) cell-based microneutralization assay (Virospot) for viruses recovered from baseline samples and viruses recovered from samples following treatment that contain amino acid changes within the MEDI8852 binding site. Participants with detectable levels (50% tissue culture infectious dose [TCID50]) of virus were considered susceptible and were reported. Due to the fact that the number of participants with viral susceptibility to MEDI8852 binding site was zero across all participant samples analyzed, no additional per arm analyses were performed.
Time Frame: From Baseline (Day 1) to Day 13
Population: PP population. Participants without confirmed influenza A at baseline were excluded from the PP population. Participants with quantifiable Influenza A (greater than LLOQ) and a unique hemagglutinin gene sequence were analyzed.
Measure: Count of Participants; unit: Participants
Groups:
- All MEDI8852 Participants: Participants who received a single IV infusion of MEDI8852 750 mg on Day 1 and oseltamivir 75 mg capsules orally BID from Day 1 to Day 5; or a single IV infusion of MEDI8852 3000 mg on Day 1 and oseltamivir 75 mg capsules orally BID from Day 1 to Day 5; or a single IV infusion of MEDI8852 3000 mg on Day 1.
Arm/Group | All MEDI8852 Participants
Number analyzed (Participants) | 35
Participants | 0

11. Secondary Outcome: Percentage of Participants With Virus Containing Known Oseltamivir Resistance-Associated Mutations
Description: Genotypic analysis was performed to identify all amino acid changes in neuraminidase (NA) gene between each baseline (Day1) sample and the participant's corresponding last sample sequenced. Percentage of participants with virus containing known oseltamivir resistance-associated mutations (change in the NA genes) is reported. Due to the fact that the percentage of participants with virus containing known oseltamivir resistance-associated mutation was zero across all participant samples analyzed, no additional per arm analyses were performed.
Time Frame: From Baseline (Day 1) to Day 13
Population: PP population. Participants without confirmed influenza A at baseline were excluded from the PP population. Participants with confirmed Influenza A positive and Influenza A concentrations greater than the LLOQ were analyzed.
Measure: Number; unit: Percentage of Participants
Groups:
- All Oseltamivir Participants: Participants who received a single IV infusion of placebo (matched to MEDI8852) on Day 1 and oseltamivir 75 mg capsules orally BID from Day 1 to Day 5; or a single IV infusion of MEDI8852 750 mg on Day 1 and oseltamivir 75 mg capsules orally BID from Day 1 to Day 5; or a single IV infusion of MEDI8852 3,000 mg on Day 1 and oseltamivir 75 mg capsules orally BID from Day 1 to Day 5.
Arm/Group | All Oseltamivir Participants
Number analyzed (Participants) | 94
Percentage of Participants | 0

ADVERSE EVENTS:
Time Frame: Treatment-Emergent Adverse Events (TEAEs) : Day 1 (post-dose) through Day 28; Treatment-Emergent Serious Adverse Events (TESAEs) : Day 1 (post-dose) through Day 101
Description: Safety analyses were performed on the as-treated population. As-treated population included all participants who were randomized and received any portion of their protocol-specified treatment regimen.
Arm/Group | Placebo + Oseltamivir 75 mg | MEDI8852 750 mg + Oseltamivir 75 mg | MEDI8852 3000 mg + Oseltamivir 75 mg | MEDI8852 3000 mg
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/31 | 0/31 | 0/31
Serious Adverse Events (participants affected / at risk) | 1/32 | 0/31 | 1/31 | 0/31
Other Adverse Events (participants affected / at risk) | 9/32 | 11/31 | 15/31 | 12/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo + Oseltamivir 75 mg (N=32) | MEDI8852 750 mg + Oseltamivir 75 mg (N=31) | MEDI8852 3000 mg + Oseltamivir 75 mg (N=31) | MEDI8852 3000 mg (N=31)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo + Oseltamivir 75 mg (N=32) | MEDI8852 750 mg + Oseltamivir 75 mg (N=31) | MEDI8852 3000 mg + Oseltamivir 75 mg (N=31) | MEDI8852 3000 mg (N=31)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (2) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 4 (4) | 5 (5) | 2 (2)
Pharyngitis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Paraesthesia (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paraesthesia oral (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Furuncle (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Polycythaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Middle ear effusion (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Administration site thrombosis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises on-going studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.